CLINICAL TRIAL: NCT05520424
Title: An Exploratory Investigation of a Supplement to Promote Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parable (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20251
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Memory Deficits; Cognitive Change; Stress
Keywords: Focus; Memory; Attention; Stress
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Daily Supplement (Experimental): Participants will use test product daily, and complete Biomarker assessments (at 1st dose, Day 7, Day 31), as well as surveys (at 1st dose, Day 7, Day 31), and Cognitive battery Assessments (at 1st dose, Day 7, Day 31).
  Interventions: Dietary Supplement: The Daily Supplement

INTERVENTIONS:
Dietary Supplement: The Daily Supplement — The ingredient list of the product includes the following:
  400mg of curcumin (Longvida) 300mg of lemon balm extract (Cyracos) 200mg of American ginseng (Cereboost) 50mg of epigallocatechin gallate derived from green tea Organic oat milk powder Phosphatidylserine (SerinAid) (active) B6 (in the form of P5P) Folate (Quatrefolic) B12 Silica (non-active)

SUMMARY:
Providing a combination of synergistic dietary supplements, such as vitamins B6, B12, and folate, as well as curcumin, lemon balm, and American ginseng is hypothesized to promote brain health and aid with brain fog, mental clarity, ability to handle stress, mood, focus, and productivity, as well as promote overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* In good general health with no major chronic conditions (e.g., diabetes, coronary heart disease, etc.)

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Anyone currently taking other supplements
* Anyone with a known allergic reaction
* Previous head trauma
* Anyone with chronic diseases such as diabetes, coronary heart disease, or cancer.
* Any psychological, mental, or neurodevelopmental disorders
* Consumes nicotine or marijuana in any form
* Previous or current alcohol addiction
* Consume more than 10 drinks per week

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Perceived changes in mental health symptoms as measured by Questionnaires | 31 days
  Questionnaires measure perceived changes in mental health symptoms (e.g., anxiety levels, mental clarity) and stress management on a scale of 0 (low levels of mental health symptoms) to 10 (very high levels of mental health symptoms)
Perceived changes in stress management as measured by Questionnaires | 31 days
  Questionnaires measure perceived changes in stress management on a scale of 0 (poor ability to manage stress) to 10 (excellent ability to manage stress)

SECONDARY OUTCOMES:
Changes in Cognitive Functioning | 31 days
  Cognitive battery questionnaires measure executive functioning, long term memory, working memory, and attention.

OTHER OUTCOMES:
Changes in plasma/serum biomarkers associated with brain health | 31 days
  Biomarkers collected via. blood sample sent to a third party lab. The biomarkers of interest for this trial include hs-CRP, HbA1c, homocysteine, and IL-6.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, PhD, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided